CLINICAL TRIAL: NCT01925911
Title: A Phase 1, Open-Label, Single-Sequence, 2-Period Study to Evaluate the Effect of IPI-145 on Single-Dose Pharmacokinetics of Midazolam (a CYP3A Substrate) in Healthy Subjects
Brief Title: Phase 1 Study in Healthy Subjects to Evaluate the Effect of IPI-145 on the Pharmacokinetics of Midazolam
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IPI-145-10
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Phase 1; Healthy subjects; DDI; CYP3A
MeSH Terms: interventions — duvelisib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-145 — 25 mg BID Oral Capsule
Drug: Midazolam — 2 mg midazolam syrup

SUMMARY:
To evaluate the effect of IPI-145 on the pharmacokinetics of midazolam, a cytochrome P450 3A (CYP3A) substrate; to assess the safety and tolerability of IPI-145 when administered with midazolam in healthy subjects.

DETAILED DESCRIPTION:
* In Treatment Period 1, subjects will receive a single 2 mg oral dose of midazolam.
* In Treatment Period 2, on Days 2-6, the same subjects will receive twice daily (BID) oral doses of 25 mg IPI-145; on Day 6, subjects will receive the morning dose of 25 mg IPI-145 concomitantly administered with 2 mg of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women of non-childbearing potential between 18-50 years of age
* Body Mass Index (BMI): 18.0 - 32.0 kg/m2.
* In good health, determined by no clinically significant findings from clinical evaluations
* Provided written informed consent prior to any study specific procedures

Exclusion Criteria:

* Women of childbearing potential
* Evidence of clinically significant medical conditions
* History of gastrointestinal disease or surgery that may affect drug absorption
* Positive or indeterminate tuberculosis-spot test at screening
* Any active infection at the time of screening or admission
* Subjects with acute narrow-angle glaucoma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (AUC) of midazolam and 1-hydroxy-midazolam | Over 24 hours
Pharmacokinetic parameters (Cmax) of midazolam and 1-hydroxy-midazolam | Over 24 hours
Pharmacokinetic parameters (t1/2) of midazolam and 1-hydroxy-midazolam | Over 24 hours
Plasma concentrations of midazolam and 1-hydroxy-midazolam | Over 24 hours

SECONDARY OUTCOMES:
Incidence of adverse events following of administration midazolam, IPI-145 and the combination | 2 weeks
  Safety Findings

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- PRA International, Lenexa, Kansas, United States